CLINICAL TRIAL: NCT04894695
Title: Identification of Biomarkers for Lupus Nephritis Using Urine Exosomes
Brief Title: Urine Exosomes to Identify Biomarkers for LN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: urine exo-LN
Record Dates: First submitted 2021-05-15; First posted 2021-05-20 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-05

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- healthy control (HC): healthy control
  Interventions: Diagnostic Test: biomarkers detection in different groups
- Systemic Lupus Erythematosus (SLE): Systemic Lupus Erythematosus
  Interventions: Diagnostic Test: biomarkers detection in different groups
- lupus nephritis (LN): lupus nephritis
  Interventions: Diagnostic Test: biomarkers detection in different groups

INTERVENTIONS:
Diagnostic Test: biomarkers detection in different groups — Biomarkers of urine exosomes in different groups were identified by sequencing technology，then biomarkers were validated using urine samples of different groups

SUMMARY:
Urine exosomes will be extracted from patients with lupus nephritis, healthy controls, and patients with systemic lupus erythematosus without lupus nephritis. Transcriptome and/or metabonomics sequencing of exosomes will be performed to screen for molecules in the urine exosomes of patients with lupus nephritis that are significantly different from those of the other groups.

DETAILED DESCRIPTION:
Lupus nephritis is one of the most common complications of SLE, and its severity is closely related to the prognosis of SLE. The gold standard for diagnosing lupus nephritis depends on the pathological results of a kidney biopsy, which is invasive and may cause some damage to the patient. Exosomes exist in almost all types of body fluids such as serum, urine and cerebrospinal fluid, and contain a variety of genetic materials and proteins secreted by cells, such as miRNA, lnRNA, cirRNA and metabolites, etc., which are potential substances that can be used as biomarkers of diseases discovered in recent years. Urine exosomes are easy to obtain and have no impact on patients' health, making them suitable for study as disease biomarkers for lupus nephritis.

In this study, urine exosomes will be extracted from patients with lupus nephritis, healthy controls, and patients with systemic lupus erythematosus without lupus nephritis. Transcriptome and/or metabonomics sequencing of exosomes will be performed to screen for molecules in the urine exosomes of patients with lupus nephritis that are significantly different from those of the other groups.

ELIGIBILITY:
Inclusion Criteria:

* No history of chronic or serious diseases such as cardiovascular disease, liver disease, kidney disease, respiratory disease, blood disease, lymphatic disease, endocrine disease, immune disease, mental disease, neuromuscular disease, gastrointestinal system disease, etc.
* General health condition is good;
* Vital signs examination, physical examination, clinical laboratory examination (blood routine, urine routine, blood biochemical examination, coagulation function examination), electrocardiogram, and the results show normal or abnormal without clinical significance

Exclusion Criteria:

* Other rheumatic immune disease;
* Abnormal liver and kidney function;
* Acute and chronic infectious diseases.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-08-02 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
specific molecule levels in urine exosomes | 2 weeks
  Molecule like miRNAs were determined in urine exosomes of different groups and the following validation will determine which molecule can be served as biomarkers of lupus nephritis

CONTACTS AND LOCATIONS:
Overall Officials: Liangjing Lu, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao Y, Wei W, Liu ML. Extracellular vesicles and lupus nephritis - New insights into pathophysiology and clinical implications. J Autoimmun. 2020 Dec;115:102540. doi: 10.1016/j.jaut.2020.102540. Epub 2020 Sep 4. PMID 32893081